CLINICAL TRIAL: NCT07310303
Title: The Effect of Simulation-Based Preoperative Education on Surgical Fear and Kinesiophobia in Patients Undergoing Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Simulation-Based Preoperative Education in Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nermin Ocaktan (Other)
Responsible Party: Sponsor-Investigator, Nermin Ocaktan, PhD, Acibadem University
Organization: Acibadem University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-18-688
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Total Knee Arthroplasty; Surgical Fear and Worrying; Kinesiophobia
Keywords: Total Knee Arthroplasty; Simulation-Based Education; Preoperative Education; Surgical Fear; Kinesiophobia; Nursing Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Kinesiophobia | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either a simulation-based preoperative education group or a standard verbal education control group, with parallel comparison of outcomes between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation-Based Preoperative Education (Experimental): Participants receive simulation-based preoperative education focusing on postoperative mobilization and recovery one day before surgery.
  Interventions: Other: Simulation-Based Preoperative Education; Procedure: Total Knee Arthroplasty
- Standard Verbal Preoperative Education (Active Comparator): Participants receive routine standard verbal preoperative education according to institutional practice.
  Interventions: Other: Standard Verbal Preoperative Education; Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Other: Simulation-Based Preoperative Education — Simulation-based education provided preoperatively to prepare patients for postoperative mobilization and recovery.
  Arms: Simulation-Based Preoperative Education
Other: Standard Verbal Preoperative Education — Routine verbal preoperative education provided according to institutional standards.
  Arms: Standard Verbal Preoperative Education
Procedure: Total Knee Arthroplasty — All participants in both study arms undergo standard total knee arthroplasty performed according to institutional clinical protocols.

SUMMARY:
This randomized controlled trial aims to evaluate the effect of simulation-based preoperative education on surgical fear and kinesiophobia in patients undergoing total knee arthroplasty. Eligible patients are randomly assigned to either a simulation-based education group or a standard verbal education (control) group. Surgical fear, kinesiophobia, and postoperative pain are assessed using validated measurement tools. The findings of this study are expected to contribute to evidence-based nursing practices by informing the development of effective preoperative education strategies to improve postoperative recovery outcomes.

DETAILED DESCRIPTION:
Total knee arthroplasty is a major orthopedic surgical procedure that may lead to significant physical and psychological challenges for patients during the perioperative period. In addition to postoperative pain and functional limitations, patients frequently experience surgical fear and fear of movement (kinesiophobia), which may negatively affect early mobilization and recovery. Preoperative education is considered an essential nursing intervention to support patients in coping with these challenges; however, the optimal method for delivering such education remains an area of ongoing research.

Simulation-based education has increasingly been used in healthcare education to enhance understanding, reduce uncertainty, and improve preparedness by allowing individuals to actively engage with the anticipated care process. While its effectiveness has been well documented in student education, evidence regarding its use in preoperative patient education, particularly in orthopedic surgery, is limited.

This randomized controlled trial aims to examine the effect of simulation-based preoperative education on surgical fear and kinesiophobia in patients undergoing primary total knee arthroplasty. Eligible patients are randomly assigned to either an intervention group receiving simulation-based preoperative education or a control group receiving standard verbal preoperative education according to institutional routine practice. The educational intervention is delivered one day prior to surgery.

Data are collected using validated instruments, including the Surgical Fear Questionnaire, the Tampa Scale of Kinesiophobia, and the Visual Analog Scale for pain assessment. Surgical fear is assessed during the preoperative period, while kinesiophobia and postoperative pain are evaluated following surgery during the early mobilization phase.

The results of this study are expected to provide evidence to inform nursing-led preoperative education strategies and to support the development of patient-centered approaches aimed at improving psychological preparedness and postoperative recovery in individuals undergoing total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Scheduled for primary total knee arthroplasty
* Able to communicate and cooperate
* Able to speak and understand Turkish
* No diagnosed major psychiatric disorder
* No diagnosed neurological disorder
* Willing to participate and able to provide written informed consent

Exclusion Criteria:

* Revision total knee arthroplasty
* Bilateral total knee arthroplasty
* Total knee arthroplasty performed due to trauma
* Presence of neurological, traumatic, or systemic conditions that may limit mobility
* Development of postoperative surgical or prosthesis-related complications
* Development of any condition preventing postoperative mobilization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Fear | Preoperative period (one day before surgery)
  Surgical fear will be assessed using the Surgical Fear Questionnaire, a validated self-report instrument measuring short-term and long-term fear related to surgery. Surgical fear will be assessed using the Surgical Fear Questionnaire, a validated self-report instrument measuring short-term and long-term fear related to surgery. Scores range from 0 to 80, with higher scores indicating greater levels of surgical fear.

SECONDARY OUTCOMES:
Kinesiophobia | Postoperative period after recovery of cognitive function
  Kinesiophobia will be measured using the Tampa Scale of Kinesiophobia, a validated self-report scale assessing fear of movement and re-injury. Scores range from 17 to 68, with higher scores indicating greater levels of kinesiophobia.
Postoperative Pain Intensity | Early postoperative period during first mobilization
  Postoperative pain intensity will be assessed using the Visual Analog Scale (VAS). Scores range from 0 to 10, with higher scores indicating greater pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Mehmet Ali Aydinlar University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves a small sample size and includes sensitive patient-reported psychological measures. Data sharing was not included in the informed consent process, and access to the dataset is restricted in accordance with institutional and ethical regulations.